CLINICAL TRIAL: NCT05445596
Title: Advancing the Effectiveness of Functional Communication Training for Children With Intellectual and Developmental Disabilities in Schools
Brief Title: Improving Treatment for Children With Intellectual and Developmental Disabilities and Problem Behavior in Schools
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources to implement intervention
Sponsor: Western Kentucky University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-037; 5P20GM103436-22 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Problem Behavior; Intellectual Disability; Developmental Disorder
Keywords: functional communication training; problem behavior; alternatives to extinction
MeSH Terms: conditions — Problem Behavior; Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The study uses single-case experimental design to identify functional relations between independent and dependent variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCT Evaluation (Experimental): This study uses single case experimental design in which participants will serve as their own control. Each participant will receive the treatment (functional communication training) and will participate in comparison conditions to evaluate the effects of the treatment. We will evaluate the effects of functional communication training during three treatment phases: initial implementation, schedule thinning, and generalization.
  Interventions: Behavioral: Functional communication training

INTERVENTIONS:
Behavioral: Functional communication training — Functional communication training (FCT) is a behavioral approach to treating problem behavior. During FCT, children learn to use communication to access reinforcers, instead of using problem behavior.

SUMMARY:
Children with intellectual and developmental disabilities (IDDs) often engage in problem behavior, and functional communication training (FCT) is a commonly used treatment for problem behavior in clinical settings. During FCT, children learn prosocial ways to request functional reinforcers (e.g., "their way") instead of using problem behavior. For example, a child who engages in self-injury to escape math instruction may be taught to exchange a break picture card to receive a brief break from the math task as an alternative to self-injury. While the efficacy of FCT is well established, less is known about its effects in school settings when procedures are necessarily adapted for feasibility. The purpose of this investigation is to develop and evaluate methods for implementing FCT for children with IDDs in school settings. The investigators will use single case experimental design, in which each participant will serve as their own control, to address the research questions. First, the investigators will evaluate the effects of providing higher quality, longer duration reinforcement for appropriate requests relative to problem behavior (e.g., 1-minute break with a preferred activity versus 20-s break alone) during FCT compared to providing equal reinforcement for appropriate requests and problem behavior. Next, the investigators will develop a treatment extension to teach children to complete academic work to gain access to their way. The investigators will use visual cues, such as a green and red index card to teach children when it is time to work and when they may access their way. The investigators will evaluate the effects of the treatment extension on academic work completion, appropriate requests, and problem behavior. Finally, the investigators will examine how visual cues influence children's behavior when educators implement intervention across different academic activities. The investigators will measure the extent to which educators implement programmed intervention procedures to inform treatment feasibility.

ELIGIBILITY:
Inclusion Criteria:

Child Eligibility Criteria

* Preschool or elementary school students between 3-11 years old
* Has an intellectual or developmental disability
* Has a functional behavior assessment and behavior intervention plan or has been identified as needing a functional behavior assessment
* Exhibits problem behavior that occurs at least daily

Adult Eligibility Criteria

* Educator who provides direct services to the child participant

Exclusion Criteria:

Child Exclusion Criteria

* Excessive absences from school
* Problem behavior occurs less frequently than daily

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage change in problem behavior | Problem behavior will be measured through study completion, up to 6 months
  The investigators will measure the frequency of problem behavior using systematic direct observation during baseline and treatment sessions. They will transform frequency of problem behavior into responses per minute and will calculate the percentage change in problem behavior during treatment sessions relative to baseline sessions at study completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to make data available to participants upon request and to submit results for publication.
Supporting Information: Study Protocol, ICF
Time Frame: The informed consent form will be available to caregivers and educators immediately after signing the form. If requested, the study protocol will be sent to the caregiver after the study is complete. Participating educators will receive copies of the study protocol during the generalization phase of the study.
Access Criteria: Each caregiver of a child enrolled in the study and each participating educator will be eligible to receive the above documents.

DOCUMENTS (2):
  • Study Protocol (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT05445596/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT05445596/SAP_001.pdf